CLINICAL TRIAL: NCT02649374
Title: Gut Microbiome and Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Eran Hadar, Dr, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0263-15-RMC
Record Dates: First submitted 2015-12-23; First posted 2016-01-07 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gestational diabetes mellitus (No Intervention): women diagnosed with GDM during pregnancy, either treated by diet or pharmacological therapy
- No GDM, Dietary Modifications (Active Comparator): Women without GDM, will be advised and monitored for dietary, Exercise and lifestyle modifications
  Interventions: Behavioral: Dietary, Exercise and lifestyle modifications
- No GDM, free diet (No Intervention): Women without GDM, for whom diet. exercise are continued regulary without any modifications

INTERVENTIONS:
Behavioral: Dietary, Exercise and lifestyle modifications — Women without GDM will receive advise on diet, exercise and lifestyle modifications similar to what is advised to women with GDM
  Arms: No GDM, Dietary Modifications

SUMMARY:
The purpose of this study is to document the gut microbiome in the 1st, 2nd and 3rd trimester among pregnant women with gestational diabetes and non diabetic controls.

DETAILED DESCRIPTION:
The gut microbiome:

The human body is colonized by a multitude of microorganisms whose collective genome, the microbiome, complements and enhances our own genome. From this perspective, humans are "supra-organisms" colonized by a number of microbial cells that is 10 times greater than the sum of all our human somatic and germ cells, and carrying 150 times more genetic information. The intestine contains the largest collection of microbes among all of our body's "habitats". In the colon, for example, bacteria reach densities of 1011 cells per gram of luminal contents. Together, gut microbes form a community, or microbiota, that has a major impact on health through interactions with host cells (including components of the innate and adaptive immune systems), through extraction of nutrients and energy from the diet, and through complex biotransformations of a variety of ingested compounds, including potential carcinogens. One of the main measures tested when analyzing bacterial populations is diversity - identifying the different microbial components in the population, and describing how similar they are to one another (according to phylogeny) both within a sample and between samples.

Changes in the gut microbiome: The majority of gut microbes are generally viewed as beneficial symbionts, but recent work has revealed that the wrong combination of beneficial microbes can be harmful. Shifts in the composition of the microbiome occur at different stages in life, such as childhood, aging, and pregnancy. Changes in the composition (dysbiosis) are also associated with a growing list of diseases, such as obesity, inflammatory bowel disease (IBD), diabetes, metabolic syndrome and others. Such associations raise the question of whether the dysbiosis contributes to, or is, a symptom of the disease. Microbiome transplant experiments have demonstrated a role of the microbiome in several diseases: several phenotypes could be transferred via the microbiota, such as enhanced fat gain, metabolic syndrome, colitis and recently, fecal transplantation from lean human subjects to human subjects with metabolic syndrome was shown to increase insulin sensitivity. Fecal transplantations have also been used successfully to treat IBD patients. Together these transplantation-based studies imply that the specific composition of the microbiota can be an important factor in the onset, and possibly the progression of chronic diseases. Thus, the gut microbiota may be considered, by extension, a factor in host fitness.

Diet and the microbiome: One of the factors that most influences the composition of the microbiome is diet. Changes in diet influence the relative abundance and composition of the microbiota almost immediately, but for these compositional changes to become stable, the dietary change has to be long term. A few examples of recent studies on how the diet impacts the microbiota are mentioned below. In humans, an increase in the ratio of Bacteroidetes/Firmicutes is observed when restricting the calorie/carbohydrate content. Reduced dietary intake of carbohydrates has also been shown to result in decreased concentrations of butyrate producing bacteria. The type and quantity of dietary fat and carbohydrate have also been shown to alter the gut microbiome of people with metabolic syndrome. Other bacteria, Prevotella for example, are associated with high intake of carbohydrates and simple sugars.

A diet high in fiber has been shown to be associated with an increase in Bifidobacterium, Lactobacillus, Enterococcus and Ruminococcus. Ruminococcus was also shown to increase in abundance in subjects on a resistant starch diet. Changes due to diet have also been described in mice. For example, a high fat diet can profoundly alter the composition of the microbiota towards an enrichment of Firmicutes.

The female microbiome: Women go through several major physiological transitions during their lifetime, beginning with puberty, followed by conception, pregnancy and finally menopause. During these changes the female body undergoes hormonal, metabolic, immunological changes, and changes in the microbiome.In a pioneering study the investigators recently showed that gut microbiota is profoundly altered in pregnancy (and changes dramatically during gestation) as compared to that in non-pregnant women. Together with what the investigators know about changes in the female vaginal microbiome (reduced microbial richness and diversity in pregnancy along with an enrichment of Lactobacilli) and other microbial changes that are unique to women (such as dramatic shifts in hormonal levels) - ] the investigators expect that different pathologies will be correlated with alterations in the microbiome.

In the proposed research, the investigators aim to test whether there is a correlation between gestational diabetes melitus and changes in the microbiome, as well as when the changes started and how glucose balance with diet changes will alter the microbiome.

The aims of the study:

1. To find out the differences in the microbiome composition between trimesters in healthy pregnant women
2. To find out the differences in the microbiome composition between GDM and healthy pregnant women during all trimesters
3. To find out the differences in the microbiome composition between balanced sugar GDM with diet and healthy women (without GDM) from GDM diagnosis till third trimester

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women at the 1st trimester

Exclusion Criteria:

1. Type 1 Diabetes Mellitus
2. Type 2 Diabetes Mellitus
3. Post Bariatric surgery
4. Any concurrent chronic illness or medication use
5. Any use of hormones or antibiotics within prior 3 months
6. Multiple gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Bacterial population diversity | 9 months
  It is a descriptive outcome descibint the physiological composition of the gut and oral microbiome. The microbiome population will be quantified by DNA analysis of the samples collected throughout pregnancy from the oral cavity and stool . The precentage of each baceria colonizing the gut and oral cavitiy will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Eran Hadar, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No